CLINICAL TRIAL: NCT00235872
Title: Open-Label Continuous Administration Study With Adalimumab (D2E7) in Subjects With Rheumatoid Arthritis
Brief Title: Adalimumab in Adult Japanese Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Abbott Japan Co.,Ltd (Industry); Eisai Co., Ltd. (Industry)
Responsible Party: Eiichi Makino, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M03-651
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Results first posted 2010-01-13 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab 40 mg every other week (eow) (Experimental)
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — 40 mg eow, sc
  Other Names: ABT-D2E7; Humira

SUMMARY:
The purpose of the study is to assess the long-term safety and tolerability of repeated administration of adalimumab in Japanese subjects with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Participation and completion until Week 24 of the prior adalimumab dose-ranging study.
* Females must be postmenopausal for at least 1 year, surgically sterile, or practicing birth control throughout the study and for 90 days after study completion.
* Female subjects tested negative in pregnancy test (serum test) at Week 24 in prior adalimumab study, if capable of pregnancy.

Exclusion Criteria:

* A subject who experienced any of the following during prior study:

  * Advanced or poorly controlled diabetes
  * Joint surgery (joint evaluated in this study)
* A subject who has been prescribed excluded medications during prior study.
* History of following during prior study:

  * Clinically significant drug or alcohol abuse
  * Intravenous (iv) drug abuse
  * Active infection with listeria or tuberculosis (TB)
  * Lymphoma, leukemia
  * And, any malignancy with the exception of successfully treated non-metastatic basal cell carcinoma of the skin.
* A subject who has been administered a live vaccine during prior study, or subject scheduled to complete the administration of a live vaccine during the study period

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2004-08; Primary Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shigeki Hashimoto, Ph.D., Study Director — Abbott
Locations (25):
- Japan (25):
  - Tokyo, Metropolis
  - Aichi, Prefecture
  - Chiba, Prefecture
  - Ehime, Prefecture
  - Fukui, Prefecture
  - Fukuoka, Prefecture
  - Gunma, Prefecture
  - Hokkaido, Prefecture
  - Hyōgo, Prefecture
  - Ibaraki, Prefecture
  - Ishikawa, Prefecture
  - Kagoshima, Prefecture
  - Kanagawa, Prefecture
  - Kyoto, Prefecture
  - Miyagi, Prefecture
  - Nagano, Prefecture
  - Nagasaki, Prefecture
  - Niigata, Prefecture
  - Okayama, Prefecture
  - Osaka, Prefecture
  - Saitama, Prefecture
  - Shizuoka, Prefecture
  - Tochigi, Prefecture
  - Tokushima, Prefecture
  - Toyama, Prefecture

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab 40 mg Eow: Adalimumab 40 mg subcutaneously (sc) administered every other week (eow) until approval of adalimumab in Japan
Period: Overall Study
Arm/Group | Adalimumab 40 mg Eow
Started | 309
Completed | 162
Not Completed | 147
Not completed — Adverse Event | 34
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 50
Not completed — Administrative reason | 61

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 309
Age, Customized [Number; unit: participants]
  < 40 years | 35
  Between 40 and 49 years | 57
  Between 50 and 59 years | 111
  >/= 60 years | 106
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 249
  Male | 60
Region of Enrollment [Number; unit: participants]
  Japan | 309

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With American College of Rheumatology (ACR) Criteria Improvement Consisting of 20%, 50%, and 70% (ACR20/50/70 Responders, Respectively)
Description: Number of responders with ACR criteria improvement consisting of 20%, 50%, and 70% (ACR20/50/70, respectively) reduction in tender or swollen joint counts (TJC or SJC, respectively) and 20%, 50%, and 70% improvement, respectively, in 3 of the following 5 criteria: 1) physician's global assessment of disease activity (PGA), 2) subject's assessment of disease activity, 3) subject's assessment of pain, 4) subject's assessment of functional disability via a health assessment questionnaire (DI-HAQ), and 5) C-reactive protein (CRP) at each visit.
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until Study completion or discontinuation (final value)
Population: Full Analysis Set - all subjects who received at least one treatment with the study drug were included in the maximum population for analysis. In this study, the safety set was defined to be identical to the full analysis set. Analysis was based on observed data.
Measure: Number; unit: participants
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 309
participants
  Week 0 ACR20 | 104
  Week 0 ACR50 | 52
  Week 0 ACR70 | 22
  Week 4 ACR20 | 157
  Week 4 ACR50 | 74
  Week 4 ACR70 | 30
  Week 8 ACR20 | 154
  Week 8 ACR50 | 74
  Week 8 ACR70 | 40
  Week 12 ACR20 | 154
  Week 12 ACR50 | 83
  Week 12 ACR70 | 39
  Week 16 ACR20 | 148
  Week 16 ACR50 | 81
  Week 16 ACR70 | 46
  Week 20 ACR20 | 155
  Week 20 ACR50 | 77
  Week 20 ACR70 | 46
  Week 24 ACR20 | 155
  Week 24 ACR50 | 91
  Week 24 ACR70 | 46
  Week 36 ACR20 | 163
  Week 36 ACR50 | 99
  Week 36 ACR70 | 50
  Week 48 ACR20 | 158
  Week 48 ACR50 | 99
  Week 48 ACR70 | 52
  Week 60 ACR20 | 141
  Week 60 ACR50 | 86
  Week 60 ACR70 | 47
  Week 72 ACR20 | 118
  Week 72 ACR50 | 75
  Week 72 ACR70 | 45
  Week 84 ACR20 | 92
  Week 84 ACR50 | 63
  Week 84 ACR70 | 33
  Week 96 ACR20 | 81
  Week 96 ACR50 | 49
  Week 96 ACR70 | 24
  Week 108 ACR20 | 72
  Week 108 ACR50 | 43
  Week 108 ACR70 | 27
  Week 120 ACR20 | 63
  Week 120 ACR50 | 41
  Week 120 ACR70 | 23
  Week 132 ACR20 | 68
  Week 132 ACR50 | 49
  Week 132 ACR70 | 27
  Week 144 ACR20 | 63
  Week 144 ACR50 | 47
  Week 144 ACR70 | 25
  Week 156 ACR20 | 61
  Week 156 ACR50 | 47
  Week 156 ACR70 | 27
  Week 168 ACR20 | 62
  Week 168 ACR50 | 42
  Week 168 ACR70 | 28
  Week 180 ACR20 | 47
  Week 180 ACR50 | 33
  Week 180 ACR70 | 16
  Week 192 ACR20 | 24
  Week 192 ACR50 | 16
  Week 192 ACR70 | 8
  Week 204 ACR20 | 8
  Week 204 ACR50 | 7
  Week 204 ACR70 | 4
  Week 216 ACR20 | 1
  Week 216 ACR50 | 1
  Week 216 ACR70 | 0
  Final Value ACR20 | 166
  Final Value ACR50 | 104
  Final Value ACR70 | 58

2. Secondary Outcome: Mean Change From Baseline in Tender Joint Count (TJC, Max=68), a Component of the American College of Rheumatology (ACR) by Visit
Description: Mean change from Baseline in TJC (max=68) at each visit, a component of ACR. For M02-575 completers, the Baseline for all efficacy analyses was defined as the Week 0 [before dosing] of the M02-575 study; for the M02-575 rescue arm, the Baseline was defined as the Week 0 [before dosing] of the M03-651 study.
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until Study completion or discontinuation (final value)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: TJC
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 309
TJC
  TJC Baseline (n=309) | 22.3 (11.59)
  TJC Week 0 (n=309) | -7.2 (10.10)
  TJC Week 4 (n=307) | -10.0 (10.10)
  TJC Week 8 (n=304) | -10.6 (10.37)
  TJC Week 12 (n=298) | -11.0 (10.70)
  TJC Week 16 (n=287) | -11.5 (10.88)
  TJC Week 20 (n=271) | -12.3 (10.84)
  TJC Week 24 (n=261) | -13.3 (10.72)
  TJC Week 36 (n=245) | -14.3 (10.43)
  TJC Week 48(n=232) | -14.9 (10.88)
  TJC Week 60 (n=209) | -15.4 (10.75)
  TJC Week 72 (n=162) | -15.9 (10.86)
  TJC Week 84 (n=125) | -16.0 (10.27)
  TJC Week 96 (n=102) | -16.0 (9.74)
  TJC Week 108 (n=95) | -16.0 (9.49)
  TJC Week 120 (n=91) | -15.9 (9.42)
  TJC Week 132 (n=90) | -16.1 (10.00)
  TJC Week 144 (n=87) | -16.4 (10.15)
  TJC Week 156(n=82) | -16.2 (11.63)
  TJC Week 168 (n=78) | -17.7 (10.43)
  TJC Week 180 (n=59) | -17.7 (11.39)
  TJC Week 192 (n=33) | -17.8 (11.75)
  TJC Week 204 (n=9) | -22.4 (8.50)
  TJC Week 216 (n=1) | -24.0 (0)
  TJC Final Value (n=309) | -12.5 (12.36)

3. Secondary Outcome: Mean Change From Baseline in Swollen Joint Count (SJC, Max=66), a Component of the American College of Rheumatology (ACR) by Visit
Description: Mean change from Baseline in SJC (max=66) at each visit, a component of ACR. For M02-575 completers, the Baseline for all efficacy analyses was defined as the Week 0 (before dosing)] of the M02-575 study; for the M02-575 rescue arm, the baseline was defined as the Week 0 (before dosing) of the M03-651 study.
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until Study completion or discontinuation (final value)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SJC
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 309
SJC
  Baseline (n=309) | 17.6 (8.26)
  Week 0 (n=309) | -6.1 (7.69)
  Week 4 (n=307) | -8.5 (7.72)
  Week 8 (n=304) | -8.6 (8.31)
  Week 12 (n=298) | -9.0 (8.09)
  Week 16 (n=287) | -9.0 (8.08)
  Week 20 (n=271) | -10.1 (7.88)
  Week 24 (n=261) | -10.9 (7.91)
  Week 36 (n=245) | -11.7 (7.83)
  Week 48 (n=232) | -11.9 (8.20)
  Week 60 (n=209) | -12.2 (8.50)
  Week 72 (n=162) | -12.8 (8.20)
  Week 84 (n=125) | -13.7 (7.73)
  Week 96 (n=102) | -13.6 (7.50)
  Week 108 (n=95) | -13.5 (7.68)
  Week 120 (n=91) | -13.8 (7.75)
  Week 132 (n=90) | -13.8 (8.17)
  Week 144 (n=87) | -14.3 (7.44)
  Week 156 (n=82) | -14.0 (7.76)
  Week 168 (n=72) | -14.7 (7.89)
  Week 180 (n=59) | -15.3 (7.76)
  Week 192 (n=33) | -17.5 (8.30)
  Week 204 (n=9) | -20.0 (4.97)
  Week 216 (n=1) | -86.0 (0)
  Final Value (n=309) | -10.6 (8.93)

4. Secondary Outcome: Mean Change From Baseline in Physician Global Assessment of Disease Activity (PGA), a Component of the ACR Criteria by Visit
Description: Change from Baseline in PGA (a visual analog scale from 0-100 mm, with 0 being the absence of disease activity and 100 mm being very strong disease activity, a component of the ACR criteria by visit). For M02-575 completers, the Baseline for all efficacy analyses was defined as the Week 0 (before dosing) of the M02-575 study; for the M02-575 rescue arm, the Baseline was defined as the Week 0 (before dosing) of the M03-651 study.
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until Study completion or discontinuation (final value).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm on a scale
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 309
mm on a scale
  Baseline (n=309) | 67.2 (19.67)
  Week 0 (n=309) | -20.0 (25.83)
  Week 4 (n=307) | -27.9 (25.80)
  Week 8 (n=304) | -28.1 (26.69)
  Week 12 (n=298) | -28.3 (26.54)
  Week 16 (n=286) | -29.9 (26.26)
  Week 20 (n=271) | -33.1 (25.59)
  Week 24 (n=261) | -35.1 (25.85)
  Week 36 (n=245) | -37.3 (24.76)
  Week 48 (n=232) | -37.8 (25.08)
  Week 60 (n=209) | -38.1 (25.75)
  Week 72 (n=162) | -39.6 (24.97)
  Week 84 (n=125) | -43.1 (23.43)
  Week 96 (n=102) | -42.8 (22.35)
  Week 108 (n=94) | -43.6 (23.47)
  Week 120 (n=91) | -42.2 (24.68)
  Week 132 (n=90) | -42.9 (24.79)
  Week 144 (n=87) | -42.3 (23.80)
  Week 156 (n=82) | -44.3 (23.73)
  Week 168 (n=78) | -45.6 (23.23)
  Week 180 (n=59) | -45.0 (26.12)
  Week 192 (n=33) | -46.1 (26.10)
  Week 204 (n=9) | -60.1 (15.52)
  Week 216 (n=1) | -64.0 (0)
  Final Value (n=309) | -30.2 (30.04)

5. Secondary Outcome: Mean Change From Baseline in Subject's Global Assessment of Disease Activity Using a Visual Analog Scale, a Component of the ACR Criteria by Visit
Description: Change from Baseline in Subject's Global Assessment of Disease Activity (a visual analog scale from 0-100 mm (0 being absence of disease activity and 100 being very strong disease activity), a component of the ACR criteria by visit). For M02-575 completers, the Baseline for all efficacy analyses was defined as the Week 0 (before dosing) of the M02-575 study; for the M02-575 rescue arm, the Baseline was defined as the Week 0 (before dosing) of the M03-651 study.
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until Study completion or discontinuation (final value).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm on unit scale
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 309
mm on unit scale
  Baseline (n=309) | 63.5 (24.00)
  Week 0 (n=309) | -14.2 (26.93)
  Week 4 (n=307) | -19.4 (28.30)
  Week 8 (n=304) | -19.8 (28.22)
  Week 12 (n=298) | -21.1 (28.62)
  Week 16 (n=287) | -21.0 (28.63)
  Week 20 (n=271) | -23.0 (29.14)
  Week 24 (n=261) | -23.9 (29.06)
  Week 36 (n=244) | -26.9 (29.38)
  Week 48 (n=231) | -27.3 (28.77)
  Week 60 (n=209) | -28.2 (29.86)
  Week 72 (n=162) | -29.4 (27.90)
  Week 84 (n=125) | -30.4 (29.49)
  Week 96 (n=102) | -31.7 (25.73)
  Week 108 (n=95) | -28.0 (27.73)
  Week 120 (n=90) | -27.9 (26.64)
  Week 132 (n=90) | -29.2 (27.73)
  Week 144 (n=87) | -28.6 (29.54)
  Week 156 (n=82) | -29.7 (28.72)
  Week 168 (n=78) | -29.7 (30.14)
  Week 180 (n=59) | -30.1 (30.45)
  Week 192 (n=33) | -22.3 (32.92)
  Week 204 (n=8) | -48.1 (30.98)
  Week 216 (n=1) | -85.0 (0)
  Final Value (n=309) | -20.7 (31.77)

6. Secondary Outcome: Mean Change From Baseline in Subject's Assessment of Pain Using a Visual Analog Scale, a Component of the ACR Criteria by Visit
Description: Change from Baseline in subject's assessment of pain (a visual analog scale from 0-100 mm [0 being no pain and 100 being unbearable pain], a component of the ACR criteria by visit). For M02-575 completers, the Baseline for all efficacy analyses was defined as the Week 0 (before dosing) of the M02-575 study; for the M02-575 rescue arm, the Baseline was defined as the Week 0 (before dosing) of the M03-651 study.
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until Study completion or discontinuation (final value).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm on unit scale
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 309
mm on unit scale
  Baseline (n=309) | 61.3 (24.03)
  Week 0 (n=309) | -12.3 (27.64)
  Week 4 (n=307) | -17.0 (28.65)
  Week 8 (n=304) | -17.7 (27.78)
  Week 12 (n=298) | -19.1 (27.66)
  Week 16 (n=287) | -19.6 (27.42)
  Week 20 (n=271) | -22.2 (27.87)
  Week 24 (n=261) | -22.7 (27.00)
  Week 36 (n=244) | -26.0 (27.55)
  Week 48 (n=231) | -26.5 (28.11)
  Week 60 (n=209) | -27.1 (28.53)
  Week 72 (n=162) | -28.6 (26.56)
  Week 84 (n=125) | -28.1 (28.65)
  Week 96 (n=102) | -30.0 (24.27)
  Week 108 (n=95) | -28.6 (24.40)
  Week 120 (n=90) | -26.3 (25.26)
  Week 132 (n=90) | -28.5 (27.13)
  Week 144 (n=87) | -27.6 (27.98)
  Week 156 (n=82) | -29.7 (26.65)
  Week 168 (n=78) | -29.4 (27.62)
  Week 180 (n=59) | -29.9 (25.63)
  Week 192 (n=33) | -23.5 (29.13)
  Week 204 (n=9) | -39.7 (30.54)
  Week 216 (n=1) | -86.0 (0)
  Final Value (n=309) | -20.1 (31.24)

7. Secondary Outcome: Mean Change From Baseline in the Disability Index of the Health Assessment Questionaire (DI-HAQ, a Component of the American College of Rheumatology (ACR) Criteria by Visit
Description: Mean change from Baseline in DI-HAQ overall score (includes 20 questions assessing physical function in 8 domains - dressing, rising, eating, walking, hygiene, reach, grip, and usual activities). Each question is on a scale of 0-3 mm to measure the ability to perform certain activities (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do so), a component of the ACR criteria by visit. DI-HAQ is derived based on the mean of individual responses not the total of individual questions
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until Study completion or discontinuation (final value)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm on a scale
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 309
mm on a scale
  Baseline (n=309) | 1.5 (0.75)
  Week 0 (n=309) | -0.2 (0.49)
  Week 4 (n=307) | -0.3 (0.53)
  Week 8 (n=304) | -0.3 (0.51)
  Week 12 (n=298) | -0.3 (0.53)
  Week 16 (n=287) | -0.3 (0.54)
  Week 20 (n=271) | -0.3 (0.56)
  Week 24 (n=261) | -0.4 (0.53)
  Week 36 (n=244) | -0.4 (0.58)
  Week 48 (n=231) | -0.4 (0.56)
  Week 60 (n=209) | -0.5 (0.57)
  Week 72 (n=162) | -0.5 (0.52)
  Week 84 (n=125) | -0.5 (0.59)
  Week 96 (n=102) | -0.5 (0.58)
  Week 108 (n=95) | -0.5 (0.55)
  Week 120 (n=90) | -0.4 (0.62)
  Week 132 (n=90) | -0.5 (0.58)
  Week 144 (n=87) | -0.5 (0.57)
  Week 156 (n=82) | -0.5 (0.58)
  Week 168 (n=78) | -0.6 (0.56)
  Week 180 (n=59) | -0.5 (0.59)
  Week 192 (n=33) | -0.5 (0.55)
  Week 204 (n=9) | -0.7 (0.48)
  Week 216 (n=1) | -1.4 (0)
  Final Visit (n=309) | -0.3 (0.62)

8. Secondary Outcome: Mean Change From Baseline in C-reactive Protein (CRP), a Component of the American College of Rheumatology (ACR) Criteria by Visit
Description: Mean change from Baseline in CRP (mg/dL), a component of the ACR criteria by visit. For M02-575 completers, the Baseline for all efficacy analyses was defined as the Week 0 [before dosing] of the M02-575 study; for the M02-575 rescue arm, the Baseline was defined as the Week 0 [before dosing] of the M03-651 study.
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until Study completion or discontinuation (final value)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 309
mg/dL
  Baseline (n=-309) | 4.7 (3.30)
  Week 0 (n=309) | -1.2 (3.02)
  Week 4 (n=307) | -1.7 (3.38)
  Week 8 (n=303) | -1.6 (3.69)
  Week 12 (n=298) | -1.5 (3.33)
  Week 16 (n=287) | -1.6 (3.58)
  Week 20 (n=271) | -1.8 (3.60)
  Week 24 (n=261) | -1.9 (3.51)
  Week 36 (n=245) | -2.2 (3.55)
  Week 48 (n=231) | -2.3 (3.66)
  Week 60 (n=209) | -2.5 (3.46)
  Week 72 (n=162) | -2.4 (3.77)
  Week 84 (n=125) | -2.9 (3.90)
  Week 96 (n=102) | -3.3 (3.59)
  Week 108 (n=95) | -3.1 (3.63)
  Week 120 (n=91) | -2.7 (4.02)
  Week 132 (n=90) | -3.3 (3.45)
  Week 144 (n=87) | -3.3 (3.37)
  Week 156 (n=82) | -3.5 (3.57)
  Week 168 (n=78) | -3.4 (3.89)
  Week 180 (n=58) | -3.2 (4.55)
  Week 192 (n=33) | -4.2 (4.21)
  Week 204 (n=9) | -5.4 (6.38)
  Week 216 (n=1) | -4.0 (0)
  Final Value (n=309) | -1.7 (4.01)

9. Secondary Outcome: Presence of Morning Stiffness
Description: The number of subjects with morning stiffness at each visit. For M02-575 completers, the Baseline for all efficacy analyses was defined as the Week 0 [before dosing] of the M02-575 study; for the M02-575 rescue arm, the Baseline was defined as the Week 0 [before dosing] of the M03-651 study.
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until Study completion or discontinuation (final value)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 309
participants
  Week 0 | 182
  Week 4 | 173
  Week 8 | 168
  Week 12 | 167
  Week 16 | 154
  Week 20 | 148
  Week 24 | 138
  Week 36 | 106
  Week 48 | 93
  Week 60 | 91
  Week 72 | 68
  Week 84 | 47
  Week 96 | 39
  Week 108 | 29
  Week 120 | 29
  Week 132 | 29
  Week 144 | 32
  Week 156 | 20
  Week 168 | 19
  Week 180 | 16
  Week 192 | 11
  Week 204 | 1
  Week 216 | 0
  Final Value | 141

10. Secondary Outcome: Mean Change From Baseline in the Duration (Minutes) of Morning Stiffness by Visit
Description: Mean change (minutes) from Baseline in morning stiffness (duration). For M02-575 completers, the Baseline for all efficacy analyses was defined as the Week 0 [before dosing] of the M02-575 study; for the M02-575 rescue arm, the Baseline was defined as the Week 0 [before dosing] of the M03-651 study.
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until Study completion or discontinuation (final value)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 309
minutes
  Baseline (n=246) | 221.8 (374.72)
  Week 0 (n=182) | -48.9 (292.93)
  Week 4 (n=173) | -64.2 (307.03)
  Week 8 (n=168) | -69.4 (387.21)
  Week 12 (n=167) | -79.7 (348.20)
  Week 16 (n=154) | -64.0 (338.37)
  Week 20 (n=148) | -87.9 (318.04)
  Week 24 (n=138) | -104.9 (293.66)
  Week 36 (n=106) | -79.9 (287.89)
  Week 48 (n=93) | -86.5 (281.83)
  Week 60 (n=91) | -95.0 (363.90)
  Week 72 (n=68) | -86.4 (247.30)
  Week 84 (n=47) | -30.5 (145.23)
  Week 96 (n=39) | -95.6 (248.27)
  Week 108 (n=29) | -97.4 (263.44)
  Week 120 (n=29) | -94.8 (278.36)
  Week 132 (n=29) | -116.9 (279.96)
  Week 144 (n=32) | -34.2 (372.50)
  Week 156 (n=20) | -46.3 (169.08)
  Week 168 (n=19) | -138.0 (338.26)
  Week 180 (n=16) | -98.8 (139.98)
  Week 192 (n=11) | -47.7 (113.65)
  Week 204 (n=1) | 30.0 (0)
  Final Value (n=238) | -57.9 (358.24)

11. Secondary Outcome: Presence of Rheumatoid Factor (RF)
Description: The number of subjects who were positive for rheumatoid factor (RF) at each visit. RF considered negative if <=20 IU/mL and positive if >20 IU/mL.
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until Study completion or discontinuation (final value)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 309
participants
  Week 24 | 248
  Week 48 | 191
  Week 72 | 142
  Week 96 | 92
  Week 120 | 69
  Week 144 | 66
  Week 168 | 60
  Week 192 | 31
  Week 216 | 1
  Final Value | 250

12. Secondary Outcome: Mean Change From Baseline in Rheumatoid Factor (IU/ML) by Visit
Description: Mean change from Baseline in RF (IU/mL). For M02-575 completers, the Baseline for all efficacy analyses was defined as the Week 0 [before dosing] of the M02-575 study; for the M02-575 rescue arm, the Baseline was defined as the Week 0 [before dosing] of the M03-651 study.
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until Study completion or discontinuation (final value)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 309
IU/mL
  Baseline (n=308) | 293.7 (412.95)
  Week 24 (n=308) | -37.6 (303.19)
  Week 48 (n=243) | -82.1 (322.10)
  Week 72 (n=185) | -104.2 (286.58)
  Week 96 (n=112) | -59.7 (445.83)
  Week 120 (n=93) | -101.0 (344.41)
  Week 144 (n=88) | -111.1 (374.58)
  Week 168 (n=80) | -139.1 (357.30)
  Week 192 (n=41) | -143.0 (428.18)
  Week 216 (n=4) | -76.0 (128.47)
  Fina Value (n=308) | -55.9 (338.06)

ADVERSE EVENTS:
Time Frame: Onset after first injection of study drug through 70 days after last injection for subjects who discontinued and through Week 216 for those who remained on study
Arm/Group | Adalimumab 40 mg Eow
Serious Adverse Events (participants affected / at risk) | 111/309
Other Adverse Events (participants affected / at risk) | 285/309
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg Eow (N=309)
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 1
Abscess (Infections and infestations) | 1
Anal fistula (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Arthritis bacterial (Infections and infestations) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Atlantoaxial instability (Musculoskeletal and connective tissue disorders) | 2
Atypical mycobacterial infection (Infections and infestations) | 2
Blood Beta-D-Glucan increased (Investigations) | 1
Bronchiectasis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 4
C-reactive protein increased (Investigations) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Cellulitis (Infections and infestations) | 4
Cerebral hemorrhage (Nervous system disorders) | 3
Cerebral infarction (Nervous system disorders) | 2
Cerebral ischaemia (Nervous system disorders) | 1
Cervical cord compression (Nervous system disorders) | 1
Cervical myelopathy (Nervous system disorders) | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chest discomfort (General disorders) | 1
Chest x-ray abnormal (Investigations) | 1
Chronic sinusitis (Infections and infestations) | 1
Colonic polyp (Gastrointestinal disorders) | 2
Computerised tomogram abnormal (Investigations) | 1
Congestive cardiomyopathy (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Cryptogenic organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Deafness neurosensory (Ear and labyrinth disorders) | 1
Decreased activity (Psychiatric disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Dermoid cyst of ovary (Congenital, familial and genetic disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Entertis infectious (Infections and infestations) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Infections and infestations) | 1
Foot deformity (Metabolism and nutrition disorders) | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastroenteritis (Infections and infestations) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1
Hand deformity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hepatic enzyme increased (Investigations) | 1
Herpes ophthalmic (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 4
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Injection site erythema (General disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Joint destruction (Musculoskeletal and connective tissue disorders) | 12
Lacunar infarction (Nervous system disorders) | 1
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lumbar spinal stenosis (Metabolism and nutrition disorders) | 2
Lung infection (Infections and infestations) | 1
Malaise (General disorders) | 1
Medical device complication (Injury, poisoning and procedural complications) | 1
Middle lobe syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Metabolism and nutrition disorders) | 1
Myelopathy (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Nervous system disorder (Nervous system disorders) | 1
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1
Osteoarthritis (Metabolism and nutrition disorders) | 2
Osteomyelitis (Infections and infestations) | 1
Osteonecrosis (Metabolism and nutrition disorders) | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Palpitations (Cardiac disorders) | 1
Parovarian cyst (Reproductive system and breast disorders) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Pericarditis (Cardiac disorders) | 1
Peripheral artery aneurysm (Vascular disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia (Infections and infestations) | 7
Pneumonia bacterial (Infections and infestations) | 2
Pneumonia staphylococcal (Infections and infestations) | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1
Pulmonary tuberculosis (Infections and infestations) | 2
Pyelonephritis (Infections and infestations) | 2
Pyelonephritis acute (Infections and infestations) | 3
Pyothorax (Infections and infestations) | 2
Pyrexia (General disorders) | 3
Radiculopathy (Nervous system disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Renal failure chronic (Renal and urinary disorders) | 1
Renal infarct (Renal and urinary disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 25
Rib fracture (Injury, poisoning and procedural complications) | 1
Scapula fracture (Infections and infestations) | 1
Secondary amyloidosis (Immune system disorders) | 1
Sepsis (Infections and infestations) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 5
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Splenic haemorrhage (Blood and lymphatic system disorders) | 1
Splenic infarction (Blood and lymphatic system disorders) | 1
Spondylolisthesis (Congenital, familial and genetic disorders) | 1
Staphylococcal bacteremia (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Subarachnoid hemorrhage (Nervous system disorders) | 2
Synovial cyst (Musculoskeletal and connective tissue disorders) | 4
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 4
Transient ischaemic attack (Nervous system disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vasodilatation (Vascular disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Weight decreased (Investigations) | 1
Endocarditis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg Eow (N=309)
Abdominal pain upper (Gastrointestinal disorders) | 17
Adverse drug reaction (General disorders) | 73
Anaemia (Blood and lymphatic system disorders) | 16
Antinuclear antibody positive (Investigations) | 38
Blood urine present (Investigations) | 21
Bronchitis (Infections and infestations) | 37
Constipation (Gastrointestinal disorders) | 42
Contusion (Injury, poisoning and procedural complications) | 38
Cough (Respiratory, thoracic and mediastinal disorders) | 26
DNA antibody positive (Investigations) | 50
Dental caries (Gastrointestinal disorders) | 24
Dermatitis contact (Skin and subcutaneous tissue disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 30
Dizziness (Nervous system disorders) | 17
Eczema (Skin and subcutaneous tissue disorders) | 31
Erythema (Skin and subcutaneous tissue disorders) | 26
Fall (Injury, poisoning and procedural complications) | 19
Gamma-glutamyltransferase increased (Investigations) | 17
Gastritis (Gastrointestinal disorders) | 17
Gastroenteritis (Infections and infestations) | 16
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 17
Headache (Nervous system disorders) | 33
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 16
Hypertension (Vascular disorders) | 25
Influenza (Infections and infestations) | 17
Injection site erythema (General disorders) | 30
Injection site reaction (General disorders) | 25
Insomnia (Psychiatric disorders) | 39
Iron deficiency anemia (Blood and lymphatic system disorders) | 21
Myalgia (Musculoskeletal and connective tissue disorders) | 18
Nasopharyngitis (Infections and infestations) | 139
Nausea (Gastrointestinal disorders) | 24
Oedema peripheral (General disorders) | 19
Osteoporosis (Musculoskeletal and connective tissue disorders) | 19
Pharyngitis (Infections and infestations) | 27
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 20
Productive cough (Respiratory, thoracic and mediastinal disorders) | 18
Pruritus (Skin and subcutaneous tissue disorders) | 37
Pyrexia (General disorders) | 26
Rash (Skin and subcutaneous tissue disorders) | 39
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 22
Stomatitis (Gastrointestinal disorders) | 21
Upper respiratory tract infection (Infections and infestations) | 36
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.